CLINICAL TRIAL: NCT01930890
Title: A Dose-Blinded, 2-Dose Level, Parallel-Group, Multicenter, Long-Term Extension Study to Evaluate the Long-Term Safety, Efficacy, and Immunogenicity of BIIB023 in Subjects With Lupus Nephritis
Brief Title: BIIB023 Long-Term Extension Study in Subjects With Lupus Nephritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results from pre-specified criteria in study NCT01499355 (211LE201) did not demonstrate sufficient efficacy to warrant continuation of the study
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 211LE202; 2013-000594-69 (EudraCT Number)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — BIIB023; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIIB023 3 mg/kg (Experimental): Participants will receive BIIB023 3 mg/kg IV every 4 weeks through Week 100 plus background therapy including oral steroids (prednisone or equivalent) and mycophenolate mofetil (MMF).
  Interventions: Biological: BIIB023; Drug: mycophenolate mofetil; Drug: oral corticosteroids
- BIIB023 20 mg/kg (Experimental): Participants will receive BIIB023 20 mg/kg IV every 4 weeks through Week 100 plus background therapy including oral steroids (prednisone or equivalent) and MMF.
  Interventions: Biological: BIIB023; Drug: mycophenolate mofetil; Drug: oral corticosteroids

INTERVENTIONS:
Biological: BIIB023
Drug: mycophenolate mofetil — titrated to a target daily dose of 2 g (1 g twice daily)
  Other Names: MMF, Cellcept
Drug: oral corticosteroids — oral corticosteroids (prednisone or equivalent) at a target prednisone dose of 10 mg/day

SUMMARY:
The primary objective of the study is to evaluate the long-term safety and tolerability of BIIB023 in participants with lupus nephritis (LN).

DETAILED DESCRIPTION:
This is an extension study for all participants who completed study 211LE201 (NCT01499355) through Week 52 and did not discontinue BIIB023 or placebo. Eligible participants from Study 211LE201 will be followed for up to 108 weeks.

Participants who received BIIB023 low dose or high dose in 211LE201 will continue to receive the same dosing in this study (211LE202; NCT01930890) in addition to background therapy. Participants who received placebo in 211LE201 are randomized to receive either BIIB023 low dose or high dose in addition to background therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who completed Week 52 of Study 211LE201 (NCT01499355) and did not discontinue BIIB023 or placebo study treatment.
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 6 months after their last dose of study treatment.

Key Exclusion Criteria:

* Any significant change in medical history in subjects from Study 211LE201, including laboratory tests or current clinically significant condition that, in the opinion of the Investigator, would have excluded the subjects' participation. The Investigator must re-review the subject's medical fitness for participation and consider any diseases that would preclude treatment under this protocol.
* Subjects from Study 211LE201 who discontinued BIIB023 or placebo treatment prior to Week 52 of Study 211LE201.
* Female subjects considering becoming pregnant while in the study, currently pregnant, or breast feeding.
* Unwillingness or inability to comply with the requirements of the protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen, makes the subject unsuitable for enrollment.

NOTE: Other Protocol-defined Inclusion/Exclusion Criteria May Apply.

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (32):
- United States (4):
  - Research Site, Lake Success, New York
  - Research Site, Columbus, Ohio
  - Research Site, Memphis, Tennessee
  - Research Site, El Paso, Texas
- Argentina (3):
  - Research Site, Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Research Site, San Juan, San Juan Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
- Research Site, Melbourne, Victoria, Australia
- Belgium (2):
  - Research Site, Leuven
  - Research Site, Liège
- Research Site, Cuiabá, Mato Grosso, Brazil
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Medellín
- France (2):
  - Research Site, Pessac, Gironde
  - Research Site, Paris, Paris Cedex 13
- Research Site, Shatin, Hong Kong
- Research Site, Debrecen, Hungary
- Research Site, Pisa, Pisa, Italy
- Malaysia (3):
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kuching, Sarawak
  - Research Site, Kuala Selangor
- Research Site, Cuauhtémoc, Mexico City, Mexico
- Research Site, Lima, Peru
- Philippines (2):
  - Research Site, Manila
  - Research Site, Quezon City
- Research Site, Lodz, Poland
- Research Site, Moscow, Russia
- Research Site, Suwon, Gyeonggi-do, South Korea
- Research Site, Sagunto, Valencia, Spain
- Thailand (2):
  - Research Site, Bangkoknoi, Bangkok
  - Research Site, Pathumwan, Bangkok

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (211LE201) to BIIB023 3 mg/kg (211LE202): Participants who received placebo every 4 weeks (Q4W) plus mycophenolate mofetil (MMF) and oral corticosteroids in 211LE201 and received BIIB023 3 mg/kg intavenously (IV) Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
- BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202): Participants who received BIIB023 3 mg/kg Q4W plus MMF and oral corticosteroids in 211LE201 and received BIIB023 3 mg/kg IV Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
- Placebo (211LE201) to BIIB023 20 mg/kg (211LE202): Participants who received placebo every 4 weeks (Q4W) plus MMF and oral corticosteroids in 211LE201 and received BIIB023 20 mg/kg IV Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
- BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202): Participants who received BIIB023 20 mg/kg Q4W plus MMF and oral corticosteroids in 211LE201 and received BIIB023 20 mg/kg IV Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
Period: Overall Study
Arm/Group | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202)
Started | 14 | 33 | 13 | 27
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 33 | 13 | 27
Not completed — Study Termination | 14 | 28 | 13 | 25
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Investigator Decision | 0 | 1 | 0 | 0
Not completed — Consent Withdrawn | 0 | 3 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (211LE201) to BIIB023 3 mg/kg (211LE202): Participants who received placebo every 4 weeks (Q4W) plus MMF and oral corticosteroids in 211LE201 and received BIIB023 3 mg/kg IV Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
- Total: Total of all reporting groups
Arm/Group | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202) | Total
Number analyzed (Participants) | 14 | 33 | 13 | 27 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.96) | 32.6 (8.93) | 31.5 (10.06) | 32.2 (8.23) | 32.1 (8.76)
Age, Customized [Number; unit: participants]
  18 to 19 years | 0 | 0 | 1 | 1 | 2
  20 to 29 years | 6 | 15 | 6 | 9 | 36
  30 to 39 years | 6 | 11 | 3 | 14 | 34
  40 to 49 years | 2 | 6 | 2 | 1 | 11
  50 to 55 years | 0 | 0 | 1 | 2 | 3
  > 55 years | 0 | 1 | 0 | 0 | 1
Gender [Count of Participants; unit: Participants]
  Female | 11 | 29 | 10 | 25 | 75
  Male | 3 | 4 | 3 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs with a start date on or after the first dose date in study 211LE202. AE: any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the subject at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect. An SAE may also be any other medically important event that, in the opinion of the Investigator, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above.
Time Frame: Up to Week 108
Population: The safety population was defined as all participants who received at least 1 dose of study treatment (3 or 20 mg/kg BIIB023 in Study 211LE202).
Measure: Number; unit: participants
Arm/Group | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202)
Number analyzed (Participants) | 14 | 33 | 13 | 27
participants
  Any event | 4 | 23 | 7 | 19
  Moderate or severe event | 2 | 12 | 3 | 6
  Severe event | 0 | 4 | 1 | 3
  Event related to dose-blinded treatment | 1 | 5 | 1 | 4
  Event related to MMF | 2 | 8 | 2 | 9
  Serious event | 1 | 7 | 4 | 3
  Serious event related to dose-blinded treatment | 0 | 2 | 1 | 1
  Serious event related to MMF | 0 | 3 | 1 | 2
  Fatal event | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment or Withdrew From Study Due to an AE
Description: as for outcome 1
Time Frame: Up to Week 108
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202)
Number analyzed (Participants) | 14 | 33 | 13 | 27
participants
  Discontinued treatment due to an AE | 0 | 0 | 0 | 0
  Withdrew from study due to an AE | 0 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to Week 108
Groups:
- Placebo (211LE201) to BIIB023 3 mg/kg (211LE202): Participants who received placebo Q4W plus MMF and oral corticosteroids in 211LE201 and received BIIB023 3 mg/kg IV Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
- Placebo (211LE201) to BIIB023 20 mg/kg (211LE202): Participants who received placebo every Q4W plus MMF and oral corticosteroids in 211LE201 and received BIIB023 20 mg/kg IV Q4W plus MMF and oral corticosteroids through Week 100 in 211LE202.
Arm/Group | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202)
Serious Adverse Events (participants affected / at risk) | 1/14 | 7/33 | 4/13 | 3/27
Other Adverse Events (participants affected / at risk) | 4/14 | 19/33 | 7/13 | 13/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) (N=14) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) (N=33) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) (N=13) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202) (N=27)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Aphakia (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 3 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (211LE201) to BIIB023 3 mg/kg (211LE202) (N=14) | BIIB023 3 mg/kg (211LE201) to BIIB023 3 mg/kg (211LE202) (N=33) | Placebo (211LE201) to BIIB023 20 mg/kg (211LE202) (N=13) | BIIB023 20 mg/kg (211LE201) to BIIB023 20 mg/kg (211LE202) (N=27)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Granulomatous liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 5 | 0 | 5
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Onychomycosis (Infections and infestations) | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 4 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 3 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Spleen palpable (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 4 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated based on the pre-specified, blinded futility analysis of Study 211LE201 (NCT01499355), which did not demonstrate sufficient efficacy to warrant continuation of the studies. Study was not terminated based on safety considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.